CLINICAL TRIAL: NCT01915459
Title: A Randomized, Double Blind, Multi-center, Active Drug Controlled, Phase III Clinical Trial to Compare the Safety and Efficacy of Botulax® Versus Botox® in Treatment of Post Stroke Upper Limb Spasticity
Brief Title: Phase III Study of Botulax® to Treat Post Stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-13-01
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Stroke; Spasticity
Keywords: Stroke; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin type A(Botulax®) (Experimental): Botulinum toxin type A
  Interventions: Biological: Botulinum toxin type A(Botulax®)
- Botulinum toxin type A(Botox®) (Active Comparator): Botulinum toxin type A
  Interventions: Biological: Botulinum toxin type A(Botox®)

INTERVENTIONS:
Biological: Botulinum toxin type A(Botulax®) — IM, total dose of 360 Units at wrist flexor, elbow flexor, finger flexor, and thumb flexor based on muscle tone
  Arms: Botulinum toxin type A(Botulax®)
Biological: Botulinum toxin type A(Botox®)
  Arms: Botulinum toxin type A(Botox®)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Botulax® compared to Botox® reducing upper limb muscle tone in post stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients, over 20 years of age
2. Patients with a history of stroke more than 6weeks prior to enrollment
3. Focal spasticity of wrist flexor measured with Modified Ashworth Scale (MAS) of 2 or greater at wrist and 1 or greater at least one of elbow flexor and finger flexor
4. A minimum grade of 2 or greater on the Disability Assessment Scale(DAS) for targeted one functional disability item (i.e., hygiene, dressing, pain, or limb position)
5. Patients who signed informed consent form, clearly understand the intent of the study and are able to comply with instructions to complete the entire study

Exclusion Criteria:

1. Patients with diagnosed neuromuscular disorders such as Lamber-Eaton syndrome, myasthenia gravis, or amyotrophic lateral sclerosis
2. Patients with profound atrophy of the muscle in the target limb
3. Patients with fixed joint/muscle contracture* in the target limb

   * Defined as inability to passively move the joints
4. Patients with history within 6 months or planned to have treatment with phenol or alcohol injection(chemodenervation) in the target limb
5. Patients with history within 6 months or planned to have treatment with tendon lengthening in the target limb
6. Patients who have concurrent treatment with an intrathecal baclofen
7. Patients who had received Botulinum toxin injection within the past 3 months(for cosmetic purpose is allowed)
8. Patients with concurrent or planned to take muscle relaxants and/or benzodiazepine medication (Allowed to participate if patient has consistently taken these medication from a month before screening visit and no changes in therapy are planned during the study)
9. Patients with concurrent or planned to have physical, occupational, or splinting therapy (Allowed to participate if these therapies were consistently taken from a month before screening visit and no treatment changes are planned during the study
10. Patients with a known allergy or sensitivity to the study medication or its components (Clostridium botulinum toxin type A, albumin, Sodium chloride, etc.)
11. Patients who have participated in other clinical trials 1 month prior to this study
12. Male and Female who are not willing to take any appropriate means of contraception or to have ascetic life at least 2 months after treatment
13. Patients who are not eligible for this study at the discretion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The change in MAS(Modified Ashworth Scale) grade | from baseline at week 4
  The change in MAS (Modified Ashworth Scale) grade from baseline at week 4 for wrist flexor muscle tone

SECONDARY OUTCOMES:
The change in muscle tone on MAS (Modified Ashworth Scale)for elbow, finger, and thumb flexor | from baseline at week 4
The change in muscle tone on MAS (Modified Ashworth Scale)for wrist, elbow, finger, and thumb flexor | from baseline at week 8 and 12
The change in DAS (Disability Assessment Scale) grade for the principal therapeutic target | from baseline at week 4, 8, 12
Global assessment evaluated by investigator | at week 4, 8, 12
Global assessment evaluated by patients | at week 4, 8, 12
The change in carer burden on Caregiver Burden Scale evaluated by caregiver | from baseline at week 4, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Min-ho Chun, Ph.D., Study Chair — Asan Medical Center
Locations (6):
- South Korea (6):
  - The Catholic University of Korea Incheon St. Mary's hospital, Incheon, Incheon
  - Seoul National University Hospital, Bundang, Kyunggi
  - Asan Medical Center, Seoul, Seoul
  - Chung Ang University Hospital, Seoul, Seoul
  - Gangnam Severance Hospital, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul